CLINICAL TRIAL: NCT04367181
Title: The Continuous Monitoring of Cerebral Function, Oxygen Perfusion and Consumption in Extremely Premature Newborns
Brief Title: DCS Study in Extremely Premature Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Angela Franceschini (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Maria Angela Franceschini, professor, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014P002022; 1R01HD091067-01A1 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-04-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Premature Birth; Extremely Low Birth Weight; Infant, Small for Gestational Age; Intracerebral Hemorrhage
Keywords: Near-Infrared Spectroscopy; Diffuse Correlation Spectroscopy; Cerebral Blood Flow
MeSH Terms: conditions — Premature Birth; Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Approximately 1.5% of infants born every year in the United States are born at an extremely low gestational age (ELGA <29 weeks GA). As reported in the 2015 VON database, the risk for developing any grade of intraventricular hemorrhage (IVH) in ELGA infants is about 20% and in more than 90% of these cases it occurs during the first three postnatal days. The major risk factor for IVH is the gestational age of the infant with greater immaturity being associated with the highest risk. The degree of prematurity of the infant relates to the immaturity of the vascular bed within the germinal matrix as well as challenges in the regulation of the cerebrovascular circulation. Specifically, increases, decreases and significant fluctuations in cerebral blood flow (CBF) have been shown to play important pathogenic roles in IVH. We are investigating the possibility of using a novel optical method to quantify cerebral perfusion, continuously, at the bedside in the NICU preterm population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ELGA group (Experimental): *Less than 29 weeks Gestational Age (GA) preemies (100)
  DCS monitoring will be performed for up to 72 hours starting within 2 days after birth. In a subgroup of infants, we will also perform additional measurements with aEEG and FDNIRS. At a second stage we will add Transcranial Doppler Ultrasound (TCD)
  Interventions: Device: Diffuse Correlation Spectroscopy (DCS); Device: Amplitude Integrated Electroencephalography (aEEG)

INTERVENTIONS:
Device: Diffuse Correlation Spectroscopy (DCS) — Diffuse correlation spectroscopy uses light in the near infrared spectral region to quantify non-invasively cerebral blood flow. The DCS device will be use to monitor blood flow changes over time in all ELGA enrolled babies
Device: Amplitude Integrated Electroencephalography (aEEG) — Amplitude Integrated Electroencephalography like EEG it is used clinically to monitor brain function in intensive care settings over longer periods of time. aEEG data will be correlated with CBF variation over time

SUMMARY:
The researchers are attempting to improve the cerebral monitoring of extremely low gestational age (ELGA) infants, such that in the future, real-time monitoring will be possible, to aid clinicians in management of these infants. The researchers wish to establish a new NIRS device, diffuse correlation spectroscopy (DCS), as a safe, noninvasive and informative bedside tool for assessing and monitoring brain health in ELGA infants during the first few days of life. It is hoped that this method will provide detailed information on changes in oxygen consumption and metabolism, and cerebral perfusion. This technique will have wide applicability, but for this research study, the researchers wish to focus on the effect of blood flow instabilities, intermittent hypotension and hypoxic episodes, pressure passive CBF periods, and hypoperfusion on the preterm brain during the first days of life, and the relationship with incidence of intraventricular hemorrhage (IVH). The researchers aim to recruit 100 premature infants to obtain data to:

1. Test the feasibility of NIRS-DCS to monitor cerebral activity, perfusion and oxygen consumption in extremely premature infants during the first week of life.
2. To assess if these baseline values are impacted by intermittent hypoxic episodes.
3. To assess if cerebral blood flow disturbances correlate with incidence of intraventricular hemorrhage.
4. Correlate the NIRS-DCS findings with clinical outcome at hospital discharge.

DETAILED DESCRIPTION:
Infants born at an extremely low gestational age (<29 weeks GA) (ELGA) are at risk for developing any grade of intraventricular hemorrhage (IVH). In association with IVH, ELGA infants may develop associated neuropathology including periventricular hemorrhagic infarction, post-hemorrhagic hydrocephalus and periventricular leukomalacia. Long-term neurodevelopmental outcomes depend on the severity of the hemorrhage. High-grade IVH (grade III or IV) is associated with a 50% risk for cerebral palsy and significant intellectual disability. Such disabilities have devastating and lifelong impact on affected children, the children's families and society. In more than 90% of the cases, IVH in ELGA infants occurs during the first three postnatal days. The major risk factor for IVH is the gestational age of the infant with greater immaturity being associated with the highest risk. The degree of prematurity of the infant relates to the immaturity of the vascular bed within the germinal matrix as well as challenges in the regulation of the cerebrovascular circulation. Specifically, increases, decreases and significant fluctuations in cerebral blood flow (CBF) have been shown to play important pathogenic roles in IVH. These CBF instabilities have been related to the mechanics of ventilation as well as to the severity of the infant's illness, with contributing factors of hypercarbia, hypovolemia, hypotension, restlessness, patent ductus arteriosus, and relatively high inspired oxygen concentrations. Another major contributing factor to CBF instabilities is the pressure-passive cerebral circulatory state in the unstable ELGA infants. To prevent such deleterious consequences on the developing brain of preterm infants, optimal therapeutic strategies that maintain both cardiopulmonary function and cerebrovascular stability need to be developed. The major obstacle impeding effective brain-oriented neonatal intensive care is the lack of a relevant bedside continuous monitor of cerebral blood flow.

Near-infrared spectroscopy (NIRS) is a non-invasive, non-ionizing method for monitoring and imaging of brain hemodynamics. Commercially available, FDA-approved NIRS systems provide hemoglobin concentration changes and relative hemoglobin oxygen saturation (rSO2) as a surrogate for cerebral perfusion and oxygen consumption. However currently there are no commercially available monitors, which can directly assess cerebral perfusion and oxygen consumption in preterm infants. The researchers are investigating the possibility of using a novel NIRS optical method to quantify cerebral perfusion, continuously, at the bedside in the NICU preterm population. The researchers believe the use of Diffuse Correlation Spectroscopy (DCS) as a stand-alone and in combination with frequency-domain (FD) or continuous wave (CW) NIRS will offer more robust diagnostic capabilities by directly quantifying cerebral blood flow (CBF), and cerebral oxygen metabolism (CMRO2). The researcher's preliminary efforts in animals and humans with this optical device show the potential of the technique.

Measurement Protocol Summary:

1. Start measurements within 48 hours of life, monitor for up to 72 hrs.
2. Up to 2 optical sensors will be attached with hydrogel, and affixed using either an infant hat headband or medical grade tapes.
3. Attached optical sensors will be adjusted every few hours to ensure that there is no disruption to skin integrity. Skin integrity will be assessed every time the optical sensors are moved and discussed with research nurse or nurse caring for infant
4. When available physiological parameters including heart rate, blood pressure, transcutaneous CO2 (TcCO2), cerebral oximetry and other systemic parameters from the bedside monitors will be collected to be compared to the optical data.
5. A research pulse oximeter will be attached to the baby to record arterial saturation (SpO2).
6. A small accelerometer will be attached to the optical sensor next to the optical sensor to record baby head motion.
7. In a subgroup of babies the researchers will also monitor enrolled infants with aEEG and FDNIRS. The aEEG leads are currently used in NICU for clinical care and the FDNIRS handheld probe is currently used in research. Depending on availability of the FDNIRS device and access to the infant, every 4 to 12 hrs, the researchers will perform FDNIRS measurements by using a hand-held optical sensor.

ELIGIBILITY:
* Premature infants born at <29 weeks GA and <48 hrs of age.
* No contraindication to DCS optical sensor placement on the scalp
* No major congenital anomalies,
* No Complex cyanotic congenital cardiac disease.

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of DCS CBF continuous measures in ELGA newborn | 5 years
  Test the feasibility of DCS monitoring of cerebral perfusion in extremely premature infants during the first few days of life.

SECONDARY OUTCOMES:
Correlation with intraventricular hemorrhage | 5 years
  To assess if cerebral blood flow disturbances measured with DCS correlate with incidence of intraventricular hemorrhage.
Correlation with clinical outcome | 5 years
  Correlate the DCS findings with clinical outcome at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Terrie E Inder, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: upon request and at study completion
Access Criteria: file share